CLINICAL TRIAL: NCT03112967
Title: Safety and Efficacy of Low-volume Preparation in the Elderly: Oral Sulfate Solution vs 4L PEG Dolution
Brief Title: Safety and Efficacy of Low-volume Preparation in the Elderly: Oral Sulfate Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Min Seob Kwak, Clinical associate professor, Kyung Hee University Hospital at Gangdong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016-03-021
Record Dates: First submitted 2017-03-30; First posted 2017-04-13 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Bowel Preparation
MeSH Terms: interventions — Polyethylene Glycols; Golytely

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSS(Suprep) (Experimental): Oral Sulfate solution (Suprep) in day before and split-dose regimens In the OSS arm: between 17:00 and 18:00 hours on the day before colonoscopy, subjects were instructed to pour one 180-ml bottle of the study medication into a provided 480-ml mixing cup and fill it with water and then drink the entire volume, followed by two additional 480 ml of water. At approximately 6:00 a.m. on the following morning, the subjects took the second dose of OSS by same formulation protocol.
  Interventions: Other: low-volume preparation, oral sulfate solution
- 4L PEG solution(Colyte) (Active Comparator): 4L PEG solution in day before and split-dose regimens In the 4L PEG arm: subjects had the first 2L between 18:00 and 19:00 hours (250mL every 15 minutes) in the evening before the colonoscopy. And the second 2L was given between 07:00 and 08:00 on the day of colonoscopy.
  Interventions: Other: large-volume preparation, 4L polyethylene glycol

INTERVENTIONS:
Other: low-volume preparation, oral sulfate solution — Oral Sulfate solution (Suprep) in day before and split-dose regimens In the OSS arm: between 17:00 and 18:00 hours on the day before colonoscopy, subjects were instructed to pour one 180-ml bottle of the study medication into a provided 480-ml mixing cup and fill it with water and then drink the entire volume, followed by two additional 480 ml of water. At approximately 6:00 a.m. on the following morning, the subjects took the second dose of OSS by same formulation protocol.
  Other Names: Suprep
  Arms: OSS(Suprep)
Other: large-volume preparation, 4L polyethylene glycol — 4L PEG solution in day before and split-dose regimens In the 4L PEG arm: subjects had the first 2L between 18:00 and 19:00 hours (250mL every 15 minutes) in the evening before the colonoscopy. And the second 2L was given between 07:00 and 08:00 on the day of colonoscopy.
  Other Names: Colyte
  Arms: 4L PEG solution(Colyte)

SUMMARY:
The investigators will investigate the safety and efficacy of low-volume preparation (Oral Sulfate solution) compared to 4L PEG solution in bowel preparation before colonoscopy.

One aim of this study was to investigate the efficacy of low-volume preparation (Oral Sulfate solution) on bowel preparation before colonoscopy.

DETAILED DESCRIPTION:
Traditionally, polyethylene glycol (PEG) solution, which requires ingestion of a large volume of liquid, has been used and now to a low-volume preparations because of its clear advantages in tolerability. The tolerability of bowel preparations is related to their volume, taste, and side effects, with this being a particular problem in the elderly. Meanwhile, a new oral sulfate solution (OSS, SUPREP, Braintree Laboratories, Braintree, Mass) formulation as an effective low-volume bowel cleansing agent, with a split-dose regimen was recently developed in 2009.

Concerned about being able to better complete ingestion of bowel cleansing agent, OSS with lower volume and improved taste features, as long as it does not sacrifice safety, shuld be a better choice than PEG. Many studies have already looked at the efficacy and safety of OSS compared to PEG in average risk population, but there are no data available in solely at the elderly population. In this context, we hypothesized that OSS could be a good alternative to a standard 4L-PEG solution in elderly patients.

In this report, we describe a multicenter, prospective, investigator-blind, randomized, controlled trial investigating OSS with 4L PEG for efficacy and safety in the elderly.

ELIGIBILITY:
Inclusion Criteria:

All participants from 65 to 75 age

Exclusion Criteria:

1. Underwent Colorectal surgery
2. CHF, Acute MI <6 months
3. ASA class III =<
4. LC, CRF, Ascite, IBD, or Severe inflammatory state
5. Severe constipation (Bowel movement 3/wk > or Taking stool softener)
6. Disabled person physically or mentally
7. Refuse consent

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 193 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-08-13 (Actual); Study Completion 2017-08-13 (Actual)

PRIMARY OUTCOMES:
Efficacy in bowel preparation | Up to 2 months
  The boston bowel preparation scale The BBPS uses a 10-point (0-9) summation scale assessing bowel preparation quality, by a 3 point scoring system of 0 to 3 in 3 segments of the colon (right colon, transverse colon, and left colon), where 0 = ''unprepared colon with mucosa not seen because of solid stool,'' 1 = ''portion of colonic mucosa of the segment seen, but other areas not well seen due to staining, residual stool, and/or opaque liquid,'' 2 = ''minor amount of residual staining, stool, and/or opaque liquid, but colonic mucosa of the segment seen well,'' and 3 = ''entire colonic mucosa seen well with no residual staining, stool or opaque liquid.'' An adequate bowel preparation was defined by a total BBPS score ≥ 6 with all segment scores ≥ 2, and excellent cleansing was considered as a score of > 7.

SECONDARY OUTCOMES:
Adverse events | Up to 2 months
  Proportion of adverse events. Adverse events recorded on the questionnaires included nausea, vomiting, abdominal pain, bloating, sleep disturbance, numbness, weakness/faint feeling, fecal incontinence, and thirsty.
  Blood samples were taken at the screening visit and the day of the procedure and were analysed for serum electrolytes (sodium, potassium, chloride, calcium, phosphate and magnesium), blood urea nitrogen (BUN), creatinine and glomerular filtration rate (GFR). Incident kidney injury was defined as a 25% increase in serum creatinine levels or longitudinal significant change in estimated glomerular filtration rate.
compliance and acceptability | Up to 2 months
  proportion of patients willingness

CONTACTS AND LOCATIONS:
Overall Officials: Min Seob Kwak, MD,PhD, Principal Investigator — KyungHee university hospital at Gangdong
Locations (1):
- Department of Internal Medicine, Kyung Hee University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Will not share datas

REFERENCES:
- [Derived] Kwak MS, Cha JM, Yang HJ, Park DI, Kim KO, Lee J, Shin JE, Joo YE, Park J, Byeon JS, Kim HG. Safety and Efficacy of Low-Volume Preparation in the Elderly: Oral Sulfate Solution on the Day before and Split-Dose Regimens (SEE SAFE) Study. Gut Liver. 2019 Mar 15;13(2):176-182. doi: 10.5009/gnl18214. PMID 30400725